CLINICAL TRIAL: NCT00719771
Title: A Multi-center Clinical Study of the Global® AP™ Shoulder in Total Shoulder Arthroplasty
Brief Title: Global® AP™ Total Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05071
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2013-12

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Glenohumeral joint; Glenoid; Shoulder arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Global® AP™ Shoulder (Other): Global® AP™ Shoulder
  Interventions: Device: Global® AP™ Total shoulder arthroplasty

INTERVENTIONS:
Device: Global® AP™ Total shoulder arthroplasty — Total shoulder arthroplasty
  Other Names: Global® AP™ Shoulder

SUMMARY:
This study will evaluate the clinical performance of DePuy Global® AP™ Shoulder prosthesis using the anchor pegged glenoid component and clinical and radiographic evaluations.

DETAILED DESCRIPTION:
The purpose of the study is to determine the difference between pre-operative and post-operative levels of patient satisfaction, shoulder function, radiographic alignment, shoulder pain and patient satisfaction in patients receiving a Global® AP™ shoulder prosthesis for glenohumeral arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected for inclusion will present for primary shoulder arthroplasty with a diagnosis of osteoarthritis and will consent to participate.

Exclusion Criteria:

* Are under 18 years of age or over 70
* Diagnosis of AVN, Inflammatory Arthritis, Fracture or Malunion.
* Have a hemi-arthroplasty
* Have destruction of the proximal humerus that precludes rigid fixation of the humeral component
* Have arthritis with insufficient cuff tissue
* Have had a failed rotator cuff surgery
* Have loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the procedure unjustified
* Have evidence of active infection
* Present with a condition of neuromuscular compromise of the shoulder (e.g., neuropathic joints or brachial plexus injury with a flail shoulder joint) - Have a known active metastatic or neoplastic disease
* Are unwilling or unable to comply with a rehabilitation program or would fail to return for the postoperative follow-up visits prescribed by the protocol
* Are skeletally immature.
* Have a known allergic reaction to implant metals, polyethylene or a tissue reaction to corrosion or wear products
* Have other conditions such as central nervous system disturbances, alcohol or drug addiction, etc. that may make effective evaluation of the joint replacement difficult or impossible
* Are currently participating in another clinical study
* Are taking > 10mg/day corticosteroids (e.g. prednisone) excluding inhalers, within 3 months prior to surgery
* Are currently involved in any personal injury litigation, medical legal or worker's compensation claims.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Constant Shoulder Score | Pre-op, 6, 12, 24 months

SECONDARY OUTCOMES:
SF-12 | Pre-op, 6,12, 24 months
Penn/ASES | Pre-Op, 6, 12, and 24 months
Radiographic Data | Pre-Op, 6 weeks, 6, 12, and 24 months
Quality of Life Survey | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sam Himden, BA, Study Director — DePuy Orthopaedics
Locations (4):
- United States (4):
  - The CORE Institute, Phoenix, Arizona
  - Mission Hospitals Research Institute, Asheville, North Carolina
  - Wellington Orthopaedics and Sports Medicine, Cincinnati, Ohio
  - Rosenberg Cooley Metcalf Clinic, Park City, Utah